CLINICAL TRIAL: NCT00545571
Title: A Single Arm, Open Label, Interventional Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Once-Monthly Administration of Intravenous C.E.R.A. for the Maintenance of Hemoglobin Levels in Hemodialysis Patients With Chronic Renal Anemia
Brief Title: MIRACLE Study: A Study of Once-Monthly Intravenous Mircera in Hemodialysis Participants With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20826
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera in Renal Anemia (Experimental): Participants will receive intravenous Mircera every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg will be determined by the dose of ESA received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within a country-specific target range.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Mircera will be administered intravenously every 4 weeks for a total of 52 weeks. The first dose of 120, 200, or 360 mcg will be determined by the dose of ESA received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within a country-specific target range.
  Other Names: Mircera

SUMMARY:
This single-arm study will assess the long-term maintenance of hemoglobin levels, safety, and tolerability of once-monthly intravenous administration of Mircera in hemodialysis participants with chronic renal anemia. Those currently receiving darbepoetin alfa, epoetin alfa, or epoetin beta maintenance treatment will receive intravenous Mircera at a starting dose of 120, 200, or 360 micrograms (mcg) per month (based on the erythropoiesis stimulating agent [ESA] dose administered on Week -1). Subsequent doses will be adjusted to maintain hemoglobin levels within the country-specific target range (11 to 13 grams per deciliter [g/dL] for Switzerland and 10 to 12 g/dL for Austria).

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Chronic renal anemia
* Hemoglobin concentration in country-specific target range (Switzerland: 11 to 13 g/dL; Austria: 10 to 12 g/dL)
* Regular long-term hemodialysis therapy with the same mode of dialysis for ≥3 months
* Continuous intravenous or subcutaneous maintenance ESA treatment during previous 2 months

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months
* Significant acute or chronic bleeding, such as overt gastrointestinal bleeding
* Active malignant disease (except non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Austria (9):
  - Bregenz
  - Feldkirch
  - Graz
  - Kufstein
  - Linz
  - Salzburg
  - Sankt Pölten
  - Steyr
  - Vienna
- Switzerland (13):
  - Basel
  - Bellinzona
  - Burgdorf
  - Geneva
  - Lausanne
  - Liestal
  - Locarno
  - Lucerne
  - Lugano
  - Mendrisio
  - Sankt Gallen
  - Sion
  - Zurich

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with erythropoiesis-stimulating agent (ESA) therapy received intravenous methoxy polyethylene glycol-epoetin beta (Mircera), also known as continuous erythropoietin receptor activator (CERA), every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 micrograms (mcg) was based upon the dose of ESA received prior to administration of study treatment, while subsequent doses were adjusted during a 16-week dose titration period (DTP) to maintain hemoglobin (Hb) concentrations within a country-specific target: 11.0 to 13.0 grams per deciliter (g/dL) in Switzerland and 10.0 to 12.0 g/dL in Austria.
Period: Overall Study
Arm/Group | Mircera in Renal Anemia
Started | 120
Completed | 53
Not Completed | 67
Not completed — Administrative Reasons | 1
Not completed — Adverse Event | 2
Not completed — Death | 5
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 2
Not completed — Refused Treatment | 1
Not completed — Screen Failure | 16
Not completed — Transfusion | 12
Not completed — Early Termination of Study | 24
Not completed — Kidney Transplantation | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of study drug and for whom data were available from at least one follow-up variable.
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with ESA therapy received intravenous Mircera/CERA, every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg was based upon the dose of ESA received prior to administration of study treatment, while subsequent doses were adjusted during a 16-week DTP to maintain Hb concentrations within a country-specific target: 11.0 to 13.0 g/dL in Switzerland and 10.0 to 12.0 g/dL in Austria.
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Average Hb Within Plus/Minus (±) 1 g/dL of Reference Hb or Within Target Range During the Efficacy Evaluation Period (EEP)
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to 0). During the EEP (Weeks 18 to 24), participants provided a total of four pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. The average Hb during the EEP was calculated per participant and assessed against the reference value. The percentage of participants who had average Hb during the EEP in the country-specific target range (11.0 to 13.0 g/dL in Switzerland and 10.0 to 12.0 g/dL in Austria) and within ±1 g/dL of their individual reference Hb was determined as the primary endpoint. The 95 percent (%) confidence interval (CI) was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: At Weeks -4, -3, -2, -1, 0; pre-dose (0 hours) and immediately before dialysis (minimum 3 sessions per week) during Weeks 18, 20, 22, 24
Population: Per Protocol (PP) Population: All participants from the Intent-to-Treat (ITT) Population who fulfill select criteria per study protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 45
percentage of participants | 75.6 [60.5 to 87.1]

2. Secondary Outcome: Mean Change in Time-Adjusted Hb From Baseline to EEP
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to 0). During the EEP (Weeks 18 to 24), participants provided a total of four pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. The average Hb during the EEP was calculated per participant and assessed against the reference value. The mean change in Hb value between reference (i.e., "Baseline") Hb and the EEP average Hb was calculated and expressed in g/dL.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 91
g/dL | -0.4 (1.09)

3. Secondary Outcome: Mean Time Spent in the Target Range for Hb During the Long-Term Safety Period (LTSP)
Description: During the LTSP (Weeks 18 to 52), participants provided a total of 16 pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. Time spent in the country-specific target range (11.0 to 13.0 g/dL in Switzerland and 10.0 to 12.0 g/dL in Austria) was defined as time from first on-target Hb to time of last known on-target Hb, as collected during the EEP. Time spent in the target range was averaged among all participants and expressed in days.
Time Frame: Pre-dose (0 hours) and immediately before dialysis (minimum 3 sessions per week) during Weeks 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40, 42, 44, 46, 48
Population: ITT Population; only participants who entered the LTSP were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 73
days | 130 (67.5)

4. Secondary Outcome: Percentage of Participants Who Maintained Average Hb Within Target Range Throughout the EEP
Description: During the EEP (Weeks 18 to 24), participants provided a total of four pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. The percentage of participants who had average Hb during the EEP in the country-specific target range (11.0 to 13.0 g/dL in Switzerland and 10.0 to 12.0 g/dL in Austria) was determined. The 95% CI was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Pre-dose (0 hours) and immediately before dialysis (minimum 3 sessions per week) during Weeks 18, 20, 22, 24
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 91
percentage of participants | 48.4 [37.7 to 59.1]

5. Secondary Outcome: Percentage of Hb Values Above or Below the Target Range During the LTSP
Description: During the LTSP (Weeks 18 to 52), participants provided a total of 16 pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. The percentage of all Hb values outside of the country-specific target range was determined and reported separately as Hb values above the upper bound (13.0 g/dL in Switzerland and 12.0 g/dL in Austria) and Hb values below the lower bound (11.0 g/dL in Switzerland and 10.0 g/dL in Austria).
Time Frame: as for outcome 3
Population: ITT Population; only those participants (n = number) who entered the LTSP and had at least one Hb excursion during the LTSP were included in the analysis.
Measure: Number; unit: percentage of Hb values
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 51
percentage of Hb values
  Above (n=32) | 22
  Below (n=51) | 38

6. Secondary Outcome: Mean Time Spent Above or Below the Target Range for Hb During the LTSP
Description: During the LTSP (Weeks 18 to 52), participants provided a total of 16 pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. Time spent outside the country-specific target range was defined as time from each off-target Hb to time of next on-target Hb, as collected during the LTSP. Time spent outside the target range was averaged among all participants and expressed in days, reported separately as time spent above the upper bound (13.0 g/dL in Switzerland and 12.0 g/dL in Austria) and time spent below the lower bound (11.0 g/dL in Switzerland and 10.0 g/dL in Austria).
Time Frame: as for outcome 3
Population: ITT Population; only those participants (n = number) who entered the LTSP and had at least one Hb excursion during the LTSP or at the last DTP visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 51
days
  Above (n=35) | 43 (45.3)
  Below (n=51) | 48 (41.2)

7. Secondary Outcome: Mean Excursions Above or Below Target Range for Hb During the LTSP
Description: During the LTSP (Weeks 18 to 52), participants provided a total of 16 pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Sampling was also performed prior to each dialysis session. Deviation from the country-specific target range was calculated as [Hb value minus country-specific upper bound] for deviations above the target range and [Hb value minus country-specific lower bound] for deviations below the target range. Deviations were averaged among all Hb values from all participants and expressed in g/dL, reported separately as mean deviation above the upper bound (13.0 g/dL in Switzerland and 12.0 g/dL in Austria) and mean deviation below the lower bound (11.0 g/dL in Switzerland and 10.0 g/dL in Austria).
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 51
g/dL
  Above (n=32) | 0.5 (0.42)
  Below (n=51) | -0.7 (0.61)

8. Secondary Outcome: Mean Number of Months a Participant Required Dose Adjustment of Mircera/CERA During the DTP and LTSP
Description: Study drug administration occurred monthly during the DTP (Weeks 0 to 16), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during Week -1. Subsequent doses could be adjusted throughout the study including during the LTSP (Weeks 18 to 52) on the basis of Hb levels or other modification criteria. The mean number of months required for dose adjustment for any reason was calculated and averaged among all participants during the DTP and LTSP.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Safety Population: All participants who received at least one dose of trial medication and at least one safety follow-up assessment, whether prematurely withdrawn or not; only those participants (n = number) who provided evaluable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 90
months
  DTP: Any Dose Change (n=90) | 1.1 (1.11)
  DTP: Dose Increase (n=90) | 0.4 (0.75)
  DTP: Dose Decrease (n=90) | 0.6 (0.87)
  LTSP: Any Dose Change (n=67) | 1.5 (1.32)
  LTSP: Dose Increase (n=67) | 0.7 (0.99)
  LTSP: Dose Decrease (n=67) | 0.8 (0.93)

9. Secondary Outcome: Mean Dose of Mircera/CERA During the DTP and LTSP
Description: Study drug administration occurred monthly during the DTP (Weeks 0 to 16), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during Week -1. Subsequent doses could be adjusted throughout the study including during the LTSP (Weeks 18 to 52) on the basis of Hb levels or other modification criteria. The dose received at each administration visit was averaged among all participants during the DTP and LTSP and expressed in mcg.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Safety Population; only those participants (n = number) who provided evaluable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 91
mcg
  DTP (n=91) | 140 (48.6)
  LTSP (n=72) | 133.8 (70.7)

10. Secondary Outcome: Percentage of Participants Who Received Blood Transfusions During the DTP and LTSP
Description: The number of participants who received blood transfusion during the DTP (Weeks 0 and 16) and LTSP (Weeks 18 to 52) was reported.
Time Frame: From Week 0 (every week until Week 2, every 2 weeks until Week 48) through the final visit at Week 52
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 91
percentage of participants | 15.4

ADVERSE EVENTS:
Time Frame: From Week -4 (every week until Week 2, every 2 weeks until Week 48) through the final visit at Week 52
Description: Safety Population.
Arm/Group | Mircera in Renal Anemia
Serious Adverse Events (participants affected / at risk) | 43/91
Other Adverse Events (participants affected / at risk) | 62/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=91)
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Pleuropericarditis (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 2
Enterococcal sepsis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Overweight (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Social problem (Social circumstances) | 1
Catheter placement (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Nephrectomy (Surgical and medical procedures) | 1
Haemodynamic instability (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=91)
Angina pectoris (Cardiac disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 7
Oedema peripheral (General disorders) | 5
Bronchitis (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 11
Fall (Injury, poisoning and procedural complications) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 12

LIMITATIONS AND CAVEATS:
The Study was prematurely terminated in Austria as a consequence of Mircera reimbursement denial. However, the Study completed regularly in Switzerland and the overall status of the Study is considered completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.